CLINICAL TRIAL: NCT07238530
Title: Evaluation of Insulin Resistance in Hepatitis C Infected Thalassemia Children and Survivors of Childhood Malignancy
Brief Title: Insulin Resistance Among Hepatitis C Infected Children
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MSO 15/2025; Pediatric Protocol (Other: Faculty of Medicine Ain Shams University)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: This Study is to Assess Occurence of Insulin Resistance Among Hepatits C Infected Children Whether Thalassemic or Survivors of Childhood Malignancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group included 60 hepatitis C infected children and adolescents: The patient group included 30 thalassemic patients and 30 malignancy survivors
- Control group of 30 age and sex matched healthy children and adolescents

SUMMARY:
The goal of this observational study was to study the occurrence of insulin resistance in hepatitis C virus infected children who were either thalassemic or survivors of childhood malignancy and its correlation to the HCV viral load and other metabolic factors.

The main question it aims to answer is:

1. Do children infected with Hepatitis C have a higher incidence of Insulin resistance compared to healthy controls of same age and gender?
2. Is Insulin resistance occurence affected by HCV viral load, blood transfusion frequency, or metabolic factors? Researchers will compare hepatitis c infected children who are either thalassemic or survivors of childhood malignant to healthy age and sex matched controls.

Participants will be subjected to:

* standardized Questionnaires,
* physical examination and
* laboratory investigations including liver functions (ALT, AST, Alkaline phosphatase), Prothrombin time, serum ferritin level, albumin, fasting glucose, fasting insulin level and Insulin resistance assessment by HOMA IR calculation.

ELIGIBILITY:
Inclusion Criteria:

* hepatitis C virus ribonucleic acid (RNA) positive children, who were following up at the pediatric hematology and oncology clinic

Exclusion Criteria:

* patients with concurrent active hepatitis B virus infection (positive for hepatitis B surface antigen) or
* autoimmune hepatitis,
* primary biliary cirrhosis (PBC),
* sclerosing cholangitis,
* haemochromatosis,
* α1-antitrypsin deficiency,
* Wilson's disease,
* patients with obesity (BMI > 25), or
* Type 2 DM.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patient group: Hepatitis C infected children and adolescents who are either thalassemia patients or survivors of childhood malignancy.
  Control group: Age and sex matched healthy children and adolescents who are following up at pediatric outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was to study the occurrence of insulin resistance in hepatitis C virus infected children who were either thalassemic or survivors of childhood malignancy | over a period of 6 months
  Insulin resistance was assessed by using Homeostasis Model Assessment (HOMA) index

SECONDARY OUTCOMES:
Secondary outcome measure was to assess correlation between insulin resistance and HCV viral load and metabolic parameters. | 6 months
  HCV viral load was measured by HCV RNA level by PCR, and metabolic parameters included liver functions, serum ferritin, fasting glucose and fasting insulin

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric hematology and Oncology clinic, Children's Hospital, Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
this study enrolled patients before January 2019